CLINICAL TRIAL: NCT00083226
Title: A Phase II Trial of Bortezomib Plus Doxorubicin in Hepatocellular Carcinoma
Brief Title: Doxorubicin and Bortezomib in Treating Patients With Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00654; NCI-2012-02952 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E6202 (Other: Eastern Cooperative Oncology Group); U10CA021115 (NIH)
Record Dates: First submitted 2004-05-14; First posted 2004-05-17 (Estimated); Results first posted 2014-10-30 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-01

CONDITIONS: Adult Primary Hepatocellular Carcinoma; Advanced Adult Primary Liver Cancer; Localized Unresectable Adult Primary Liver Cancer; Recurrent Adult Primary Liver Cancer
Keywords: doxorubicin; doxorubicin hydrochloride; bortezomib; hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Doxorubicin; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (doxorubicin+bortezomib) (Experimental): Patients receive doxorubicin IV over 5-15 minutes on days 1 and 8. Patients also receive bortezomib at a dose of 1.3 mg/m^2 IV over 3-5 seconds on days 1, 4, 8, and 11. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patients with no disease progression may continue to receive bortezomib alone in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: doxorubicin; Drug: bortezomib

INTERVENTIONS:
Drug: doxorubicin — Given IV
  Other Names: doxorubicin hydrochloride; ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE

SUMMARY:
This phase II trial is studying how well giving doxorubicin together with bortezomib works in treating patients with liver cancer. Drugs used in chemotherapy, such as doxorubicin, work in different ways to stop tumor cells from dividing so they stop growing or die. Bortezomib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Giving doxorubicin together with bortezomib may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the tumor response rate in patients with hepatocellular carcinoma (HCC).

SECONDARY OBJECTIVES:

I. To determine other parameters of antitumor effect including time to tumor progression and overall survival in HCC patients treated with bortezomib and doxorubicin.

II. To observe toxicity profile of bortezomib and doxorubicin in patients with hepatocellular carcinoma.

III. To evaluate proteasome 20S inhibition in tumor tissue (including proteins such as p21, p27, p53, Bax and Bcl-2 which are affected by proteasome 26S) and compare them to clinical parameters using biopsy specimens obtained from patients with HCC treated with bortezomib. (Withdrawn as of 03-2007)

IV. To measure phosphorylation of IkB in tumor tissue and compare to clinical parameters using biopsy specimens obtained from patients with HCC treated with bortezomib. (Withdrawn as of 03-2007)

V. To evaluate the effect of bortezomib on 26S proteasome activity in peripheral white blood cells (WBC's) and patient serum. Direct measurement of 26S proteasome activity as well as proteins affected by proteasome 26S and Nuclear factor kappa-B (NF-kB) will be analyzed. (Withdrawn as of 03-2007)

OUTLINE: This is a multicenter study.

Patients receive doxorubicin intravenously (IV) over 5-15 minutes on days 1 and 8. Patients also receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patients with no disease progression may continue to receive bortezomib alone in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 1 year.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 13 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have microscopically confirmed hepatocellular carcinoma not amenable to curative resection; if patients have an isolated lesion in one lobe of the liver, a liver surgeon should determine resectability; central review is not required
* Patients must have measurable disease as determined by Response Evaluation Criteria In Solid Tumors (RECIST) criteria, amenable to biopsy; patients are not mandated to allow biopsy, even though it is an important aspect of this clinical trial
* Patients with history of malignancy treated within the past 5 years are not eligible; history of carcinoma-in-situ of cervix, squamous cell cancer of skin, basal cell cancer of skin, previously treated are allowed; others are excluded as recurrence of disease may confuse response rate and/or survival endpoints
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Patients must not have had prior systemic chemotherapy for HCC; patients on antineoplastics for non-malignant diseases, such as methotrexate for rheumatoid arthritis, are allowed, providing patients have been off these agents for at least 4 weeks and all related toxicities have resolved to baseline
* Patients may have had prior embolization without chemotherapy; patients who have had chemoembolization are not eligible; patients may have had radiofrequency (RF) ablation, cryosurgery or ethanol injection; patients must have documented progression with the involved lesion or at least one previously untreated lesion amenable to biopsy
* Platelet count must be >= 100,000/mm^3 in absence of splenomegaly; platelet count must be >= 75,000/mm^3 with splenomegaly
* Absolute neutrophil count (ANC) must be >= 1,500/mm^3 in absence of splenomegaly; ANC must be =< 1,000/mm^3 with splenomegaly
* Alkaline phosphate (ALT) must be =< 5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) must be =< 5 x institutional ULN
* Bilirubin must be =< 2 mg/dl
* Patients may not exhibit Child Pugh scale grade C cirrhosis
* Serum creatinine=< 2.0 mg/dl
* All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy
* Women of childbearing potential and sexually active males are strongly advised to use an accepted and effective method of contraception
* Patients must not have known bleeding diathesis, international normalized ratio (INR) > 1.5 or Partial thromboplastin time (PTT) > 1.5 x institutional ULN (required due to biopsy portion of study); use of vitamin K or fresh frozen plasma to correct values just prior to biopsy or enrollment is not allowed are not eligible

Exclusion criteria:

* Patients have baseline peripheral neuropathy > grade 1
* Patients with history of untreated malignancy other than HCC
* Patients have had prior use of octreotide or tamoxifen as therapy for HCC
* Patients with known allergy to boron, mannitol or bortezomib
* Women are pregnant or breast-feeding (due to the uncertain effects of bortezomib in the developing fetus and young infants)
* Patients have an underlying medical condition that precludes safe participation in this clinical trial
* Patients have psychiatric illness or continued substance abuse that may impair the ability to provide informed consent or prevent safe administration of bortezomib
* Patients with ejection fraction (EF) < 50% measured by Echocardiography (ECHO) or Multiple gated acquisition (MUGA)
* Patients on verapamil who cannot be switched to an alternative medication (due to the interaction with doxorubicin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2004-03; Primary Completion 2011-02 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Berlin, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Ciombor KK, Feng Y, Benson AB 3rd, Su Y, Horton L, Short SP, Kauh JS, Staley C, Mulcahy M, Powell M, Amiri KI, Richmond A, Berlin J. Phase II trial of bortezomib plus doxorubicin in hepatocellular carcinoma (E6202): a trial of the Eastern Cooperative Oncology Group. Invest New Drugs. 2014 Oct;32(5):1017-27. doi: 10.1007/s10637-014-0111-8. Epub 2014 Jun 4. PMID 24890858

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on March 19, 2004 and terminated on February 12,2007 after meeting its accrual goal of 40 patients. The final accrual of the study was 42 patients, enrolled through 4 ECOG member institutions.
Groups:
- Treatment (Doxorubicin+Bortezomib): Patients receive doxorubicin IV over 5-15 minutes on days 1 and 8. Patients also receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patients with no disease progression may continue to receive bortezomib alone in the absence of disease progression or unacceptable toxicity.
  doxorubicin: Given IV
  bortezomib: Given IV
Period: Overall Study
Arm/Group | Treatment (Doxorubicin+Bortezomib)
Started | 42
Completed | 0
Not Completed | 42
Not completed — Lack of Efficacy | 19
Not completed — Adverse Event | 9
Not completed — Death | 4
Not completed — Withdrawal by Subject | 4
Not completed — Other | 2
Not completed — ineligible or not receiving treatment | 4

BASELINE CHARACTERISTICS:
Population: The primary population was the 38 eligible and treated patients
Arm/Group | Treatment (Doxorubicin+Bortezomib)
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate Measured by Response Evaluation Criteria In Solid Tumors (RECIST)
Description: Tumor response was measured by Response Evaluation Criteria In Solid Tumors (RECIST) v1.0. Objective response rate included complete response (disappearance of all tumor lesions) and partial response (At least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum longest diameter.).
Time Frame: assessed every 3 cycles while on treatment. After discontinuing treatment, assessed every 3 months for 2 years and then every 6 months for 1 year
Population: eligible and treated patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Doxorubicin+Bortezomib)
Number analyzed (Participants) | 38
percentage of participants | 3 [0.1 to 12]

2. Secondary Outcome: Overall Survival
Description: Overall survival is defined as time from registration to death from any cause. Patients alive were censored at follow up. Analysis was conducted in the 38 eligible and treated patients.
Time Frame: assessed every 3 months for 2 years and then every 6 months for 1 year
Population: eligible and treated
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Doxorubicin+Bortezomib)
Number analyzed (Participants) | 38
months | 6.4 [4.4 to 8.5]

3. Secondary Outcome: Progression Free Survival
Description: Time from registration to disease progression or death, whichever occurred earlier. Patients alive and progression-free were censored at last follow up. 36 eligible and treated patients were included in the analysis. The other 2 eligible and treated patients had no disease status information.
Time Frame: as for outcome 1
Population: eligible and treated patients with progression status information
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Doxorubicin+Bortezomib)
Number analyzed (Participants) | 36
months | 2.2 [2.0 to 3.4]

ADVERSE EVENTS:
Time Frame: Assessed every while on treatment and for 30 days after the end of treatment
Groups:
- Doxorubicin+Bortezomib: Patients receive doxorubicin IV over 5-15 minutes on days 1 and 8. Patients also receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11.
Arm/Group | Doxorubicin+Bortezomib
Serious Adverse Events (participants affected / at risk) | 28/39
Other Adverse Events (participants affected / at risk) | 36/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Doxorubicin+Bortezomib (N=39)
Anemia (Blood and lymphatic system disorders) | 2
Leukocytes decreased (Investigations) | 11
Neutrophils decreased (Investigations) | 8
Platelets decreased (Investigations) | 16
Fatigue (General disorders) | 7
Activated partial thromboplastin time pr (Investigations) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 5
Dysphagia (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Infection w/ gr3-4 neut, lung (Infections and infestations) | 1
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Abdomen, pain (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Doxorubicin+Bortezomib (N=39)
Anemia (Blood and lymphatic system disorders) | 33
Leukocytes decreased (Investigations) | 24
Neutrophils decreased (Investigations) | 16
Platelets decreased (Investigations) | 28
Fatigue (General disorders) | 22
Fever w/o neutropenia (General disorders) | 2
Insomnia (Psychiatric disorders) | 2
Weight loss (Investigations) | 4
INR increased (Investigations) | 2
Activated partial thromboplastin time pr (Investigations) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3
Pruritus/itching (Skin and subcutaneous tissue disorders) | 4
Skin-other (Skin and subcutaneous tissue disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 14
Constipation (Gastrointestinal disorders) | 9
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 11
Dyspepsia (Gastrointestinal disorders) | 3
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 14
Taste disturbance (Nervous system disorders) | 7
Vomiting (Gastrointestinal disorders) | 5
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Edema limb (General disorders) | 2
Alkaline phosphatase increased (Investigations) | 16
Aspartate aminotransferase increased (Investigations) | 24
Blood bilirubin increased (Investigations) | 10
Creatinine increased (Investigations) | 9
Hyponatremia (Metabolism and nutrition disorders) | 2
Neuropathy-sensory (Nervous system disorders) | 10
Abdomen, pain (Gastrointestinal disorders) | 5
Muscle, pain (Musculoskeletal and connective tissue disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less